CLINICAL TRIAL: NCT00210119
Title: Multicentric Phase II Study to Evaluate Feasibility and Efficacy of Association of Imatinib Mesylate and Zoledronic Acid in Patients With Chronic Myeloid Leukaemia in Cytogenetic Response Without Molecular Response After One Year of Imatinib Mesylate Monotherapy
Brief Title: Imatinib Mesylate and Zoledronic Acid in Patients With Chronic Myeloid Leukaemia in Cytogenetic Response Without Molecular Response
Acronym: AFR22
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2005-25; AFR22
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-09

CONDITIONS: Myeloid Leukemia, Chronic
Keywords: Chronic myeloid leukemia; imatinib mesylate; zoledronate; molecular response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

ARMS (1):
- Imatinib mesylate (Experimental): Imatinib mesylate 600 or 800 mg/day PO + zoledronate 4 mg IV over 15 min every 3 weeks for 6 months.
  Interventions: Drug: Glivec

INTERVENTIONS:
Drug: Glivec

SUMMARY:
Imatinib mesylate is standard treatment of Chronic myeloid leukaemia, complete cytogenetic response is obtained in most of cases but molecular response concerned only a small part of the patients. To increase molecular response ratio we decided to increase imatinib dose to limited resistance to this drug and to add zoledronate for it anti tumoral activity to increase anti leukemic effect. We plan to accrue 37 patients in 5 centers. We will analyse molecular expression of BCR-ABL transcript after 6 months of treatment, safety, duration of response, VEGF expression and LTgd production.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: at registration· Chronic myeloid leukaemia Ph+ confirmed by cytogenetic analysis or BCR-ABL translocation by molecular biology· Chronic phase:-<15% blast cells in blood and 5% in bone marrow-<30% blast cells+promyelocyte cells in blood and bone marrow-<20% basophils in blood->100.000 platelets· Without extra medullar attempt excepted hepatosplenomagalia· First line of treatment· Biology and biochemistry with normal levels· Male or female>18 years old· Signed written consent· ECOG<3At inclusion· Chronic myeloid leukaemia with cytogenetic response without molecular response after one year of treatment by imatinib and BCR-ABL transcript detected by RT-PCR

Exclusion Criteria:

* · Other cancer excepted basocellular or cervix carcinoma · Major surgery in last 2 weeks previous inclusion· Women who are pregnant or breastfeeding (are unable to use an acceptable method to avoid pregnancy of his partner for the entire study period)· Dementia or altered mental status that would prohibit the understanding or rendering of informed consent · Abnormal renal function with creatinine clearance < 30 ml/ minuteAccording to Cockcroft-Gault : CrCl= [[140-age (years)] x weight (kg)]/ [72 x serum creatinine (mg/dL)] {x 0.85 for women}· Chronic myeloid leukaemia in acute phase or in pass to be in acute phase · Treatment with bisphosphonates in last 6 months previous inclusion · Intolerance to bisphosphonates: hypersensitivity, on course dental problem, including tooth or mandibular infection; dental traumatism or recent diagnosis or previous mandibular osteonecrosis, or dental extraction with cicatrisation delay or necessity to set bone evidence · Mandibular surgery in last 6 weeks or planned in the future during treatment (tooth extraction)· Serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive protocol therapy: diabetes, thyroid pathology, neuropsychiatric illness, myocardial infarction or congestive heart failure grade 3-4 according to " New York Heart association"· History of psychiatric or depressive pathology · HIV positivity known · Inclusion in other study investigating antineoplastic molecule in last 30 days previous inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-07-12 (Actual); Primary Completion 2007-09 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josy REIFFERS, Pr, Principal Investigator — Institut Bergonié
Locations (7):
- France (7):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Institut Bergonié - Centre Régional de Luttre Contre le Cancer de Bordeaux et du Sud Ouest, Bordeaux
  - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Archet, Nice
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The AFR-22 trial was based on a two-stage Simon's design, which included 17 patients in the first stage, followed by an additional 20 patients. Analysis of the first 17 evaluable patients showed insufficient efficacy of the study treatment. In accordance with the principle of Simon's two-stage design, enrollment was stopped.
Groups:
- Imatinib Mesylate: Imatinib mesylate 600 or 800 mg/day PO + zoledronate 4 mg IV over 15 min every 3 weeks for 6 months.
  Glivec
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 19
Completed | 17
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 58.4 [32.7 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Region of Enrollment [Count of Participants; unit: Participants]
  France | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Molecular Response
Description: A patient is considered to be in molecular response if at least one of the following conditions is observed :
  - a complete molecular response at 6 months defined by PCR negativation tested on twice
  OR
  - reduction of BCR-ABL transcript level > 2 Log from the start of from initiation of treatment
Time Frame: 6 months
Population: 2 patients were not assessable for the primary outcome measure : 1 not eligible and 1 not treated because of withdrawal
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 17
percentage of participants | 0 [0 to 0]

2. Secondary Outcome: Percentage of Participants With a Reduction of BCR-ABL Transcript Level > 4.5 Log From the Start of From Initiation of Treatment
Description: reduction of BCR-ABL transcript level > 4.5 Log from the start of from initiation of treatment
Time Frame: 6 months
Population: 2 patients were not assessable for secondary outcome measures
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 17
percentage of participants | 0 [0 to 0]

ADVERSE EVENTS:
Description: Only serious adverse events were monitored. Adverse events (non-serious) were not assessed/monitored during the study.
Arm/Group | Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (N=17)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Acute pulmonary edema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes